CLINICAL TRIAL: NCT06257576
Title: Function of Tamsulosin in Older Males Undergoing Surgery with Indwelling Catheter: a Randomized Clinical Trial
Brief Title: Function of Tamsulosin in Older Males Undergoing Surgery with Indwelling Catheter
Acronym: FOLI
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: ABRAHAM J & PHYLLIS KATZ FOUNDATION (Unknown)
Responsible Party: Principal Investigator, Kenneth Cardona, Professor of Surgery, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006810
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Postoperative Urinary Tract Infection
Keywords: post-operative urinary retention (POUR); catheter-associated urinary tract infection (CAUTI); Flomax; Foley Catheter
MeSH Terms: interventions — Tamsulosin; Control Groups; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tamusolin (Experimental): Participants will receive tamsulosin postoperatively for two days.
  Interventions: Drug: Tamsulosin
- Control Group (Other): Participants will be randomized to the standard of care, with no medication given.
  Interventions: Other: Control Group

INTERVENTIONS:
Drug: Tamsulosin — Tamsulosin is a selective antagonist at alpha-1A and alpha-1B-adrenoreceptors in the prostate, prostatic capsule, prostatic urethra, and bladder neck. Blockage of the alpha-1A receptors causes relaxation of smooth muscles in the bladder neck and prostate, thus decreasing urinary outflow resistance in men.
  Tamsulosin will be administered twice a day for two (2) days as an oral tablet containing 0.4 mg of the drug. It is usually administered 30 minutes after a meal to minimize plasma level variations. The 0.4 mg dose of tamsulosin that will be used in this trial has shown adequate safety and tolerability in multiple previously published studies as well as efficacy in treating benign prostatic hyperplasia (BPH) and lower urinary tract symptoms in men.
  A Foley catheter, which will be placed for the participant's surgical procedure regardless of enrollment in the study, will be removed at midnight on postoperative day 1.
  Other Names: Flomax
  Arms: Tamusolin
Other: Control Group — A Foley catheter, which will be placed for the participant's surgical procedure regardless of enrollment in the study, will be removed at midnight on postoperative day 1.
  Other Names: Standard of Care (SOC)
  Arms: Control Group

SUMMARY:
This study is being done to answer the question: What is the impact of a medication called tamsulosin (also called Flomax) on the rate of postoperative urinary retention (POUR) and catheter-associated urinary tract infection (UTI)? One of the most common complications following surgery and associated with Foley catheters is post-operative urinary retention (POUR) after the catheter is removed. This is defined as being unable to urinate spontaneously within 8 hours following the removal of the indwelling Foley catheter (the catheter that sits in your bladder to drain urine after surgery). When this happens, it requires intermittent straight catheterization of the bladder (placing a temporary catheter in the bladder to drain the buildup of urine), which can cause a lot of discomfort and anxiety, as well as increase the risk of catheter-associated urinary tract infection (CAUTI).

DETAILED DESCRIPTION:
All participants in this study will be males who are undergoing a planned surgery on their liver, gallbladder/biliary tract, pancreas, colon, or rectum for any reason. If able to obtain appropriate consent from a legal representative, cognitively impaired patients may be included. After having surgery where a catheter is placed in the bladder to drain urine (this is called a Foley indwelling catheter), the catheter eventually gets removed, and some of the most frequent problems that can happen after that are post-operative urinary retention (POUR) and catheter-associated urinary tract infection (CAUTI).

The goal of this study is to see if a medicine called tamsulosin (also called Flomax) can decrease the rate of POUR, which means not being able to urinate spontaneously like normal, and CAUTI, which means an infection in the urinary tract. This study is important because POUR and CAUTI can cause harm to patients, including discomfort if a temporary catheter has to be placed back in the bladder to get the urine out, infection, anxiety, and stress, and it's known that these complications can also increase hospital charges.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective surgery for any reason (benign, malignant, or indeterminate lesion) with either an open or minimally invasive approach (hepatobiliary, pancreatic, and colorectal operations)
* Male and age ≥50 years
* Deemed physically fit for surgery

Exclusion Criteria:

* Inability to obtain informed consent
* Age <50 years
* Female
* Baseline creatinine >1.5x upper limit of normal
* Tamsulosin therapy as a home-medication
* Procedure involving the prostate, bladder, ureters, or kidneys
* Planned Foley catheter removal on the same day of surgery
* Planned nasogastric tube retention on postoperative day 1
* Individuals taking daily phosphodiesterase 5 (PDE5) inhibitors (due to the risk of symptomatic hypotension if given with tamsulosin)

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The investigational product (IP)Tamsulosin is used in men to treat the symptoms of an enlarged prostate (benign prostatic hyperplasia or BPH)
Enrollment: 212 (Estimated)
Dates: Start 2024-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants who develop postoperative urinary retention (POUR) postoperatively (efficacy). | Up to 3 days post-surgery
  Researchers will document the incidence of postoperative urinary retention (POUR) rate, as defined as the inability to void within 8 hours after Foley catheter removal at midnight on postoperative day 1.

SECONDARY OUTCOMES:
Number of participants with catheter-associated urinary tract infections (CAUTI), | Up to 5 days post-surgery
  Participants who develop CAUUTI, defined by positive urinary analysis (UA) or bacterial culture >100,000 colony-forming units (CFUs), within the first 5 days following surgery or until hospital discharge, whichever comes first.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Cardona, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital (EUH), Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: Yes
The Research Team will share the National Surgical Quality Improvement Program (NSQIP) de-identified data upon request.
Supporting Information: Study Protocol, SAP
Access Criteria: The Investigator will share the NSQIP de-identified data for a secondary analysis of the data upon request.